CLINICAL TRIAL: NCT00271245
Title: Selenium Supplementation of Patients With Cirrhosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds to complete study.
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, RBurk, M.D., Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK58763-c; R01DK058763 (NIH); DK58763
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Liver Disease
Keywords: cirrhosis; liver disease; selenium; selenoproteins; selenoprotein P; biomarkers
MeSH Terms: conditions — Liver Diseases; Fibrosis | interventions — Selenium; Selenic Acid; Selenomethionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 200 µg selenium as selenate
  Interventions: Dietary Supplement: 200 µg selenium as selenate
- 2 (Experimental): 400 µg selenium as selenate
  Interventions: Dietary Supplement: 400 µg selenium as selenate
- 3 (Experimental): 200 µg selenium as selenomethionine
  Interventions: Dietary Supplement: 200 µg selenium as selenomethionine
- 4 (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 200 µg selenium as selenate — 200 µg selenium as selenate
  Arms: 1
Dietary Supplement: 400 µg selenium as selenate — 400 µg selenium as selenate
  Arms: 2
Dietary Supplement: 200 µg selenium as selenomethionine — 200 µg selenium as selenomethionine
  Arms: 3
Dietary Supplement: Placebo — Placebo
  Arms: 4

SUMMARY:
The purpose of this study is to determine whether patients with liver cirrhosis can improve their selenium nutritional status by taking supplemental selenium.

DETAILED DESCRIPTION:
Selenium is an essential nutrient. Selenium carries out its biological functions through selenoproteins. The liver converts dietary selenium to a form that can be used to make selenoproteins. Patients with cirrhosis have much lower selenium levels than healthy individuals. We hypothesize that patients with cirrhosis are unable to utilize dietary selenium for selenoprotein synthesis. These patients may benefit from another form of selenium: selenate.

We will compare the effects of two supplemental forms of selenium on plasma selenium levels in patients with cirrhosis. Patients will be randomized to receive either a placebo, 200 µg selenomethionine, 200 µg selenate or 400 µg selenate, daily, for 8 weeks. We will measure selenium levels in the blood at baseline, week 4 and week 8. We will determine which forms of selenium, if any, increased plasma selenium levels of the cirrhosis patients.

ELIGIBILITY:
Inclusion Criteria:

* liver disease
* aged 18 or above

Exclusion Criteria:

* substance abuse
* renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Plasma selenoprotein P, Plasma GPX-3 activity, Total plasma selenium | 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Burk, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Burk RF, Hill KE, Motley AK, Byrne DW, Norsworthy BK. Selenium deficiency occurs in some patients with moderate-to-severe cirrhosis and can be corrected by administration of selenate but not selenomethionine: a randomized controlled trial. Am J Clin Nutr. 2015 Nov;102(5):1126-33. doi: 10.3945/ajcn.115.110932. Epub 2015 Oct 14. PMID 26468123